CLINICAL TRIAL: NCT06376903
Title: Effect of Pilates Exercises on Stress Urinary Incontinence in Posmenopausal Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eslam Mohmedy Mosa, Cairo university, Cairo University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004860
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Urinary Stress Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group ; of pilates exercises,Kegel exercises,and home care advices.advices (Active Comparator): •study group : It will be consisted of thirty postmenopausal women suffering from mild and moderate stress urinary incontinence, will perform program of pilates exercises, 3 sessions/week (30 minutes a session ) for 12 weeks in addition to Kegel exercises (15min/three times per week/ for 12 weeks) and home care advices.
  Interventions: Other: Pilates exercise - pelvic floor exercise - home advices
- Controlled group;Kegel exercises,and home care advices. (Active Comparator): Controlled group : It will be consisted of thirty postmenopausal women suffering from mild and moderate stress urinary incontinence, will perform kegel exercises (15min/three times per week/ for 12 weeks) and home care advices as in group (A).
  Interventions: Other: Pilates exercise - pelvic floor exercise - home advices

INTERVENTIONS:
Other: Pilates exercise - pelvic floor exercise - home advices — Group (A) (Study group): It will be consisted of thirty postmenopausal women suffering from mild and moderate stress urinary incontinence, will perform program of pilates exercises, 3 sessions/week (30 minutes a session ) for 12 weeks in addition to Kegel exercises (15min/three times per week/ for 12 weeks) and home care advices.
  • Group (B) (Controlled group): It will be consisted of thirty postmenopausal women suffering from mild and moderate stress urinary incontinence, will perform kegel exercises (15min/three times per week/ for 12 weeks) and home care advices as in group (A).
  Other Names: Pelvic floor exercise - home care advices

SUMMARY:
• This study will be conducted to determine the effect of pilates exercises on stress urinary incontinence in postmenopausal women

DETAILED DESCRIPTION:
Pilates exercises help in the controlled movement of the core, that act as a corset and it activates both core muscle and synergistically the PFM. (Trantafylidis, 2009).

There is limited evidence regarding the use of Pilates exercises for the management of stress urinary incontinence (SUI) in older women (Keri, 2013; Pyria et al, 2021). So this study will be conducted to determine the effect of Pilates exercises on SUI in postmenopausal women which provide an insight about the benefits of such exercise on postmenopausal SUI.

ELIGIBILITY:
Inclusion Criteria:Postmenopausal women (at least 12months after menstrual cessation), diagnosed with SUI by the gynecologist.

* Their ages will range from 50-60 years old .
* Their BMI will be less than 30kg/m2 .
* All of them suffer from mild to moderate degree of SUI .
* All of them delivered vaginally.
* All are multipara with 2 or more children.
* All are of sedentary life style.

Exclusion Criteria:Women will be excluded from the study if they have:

* Previous bladder surgery.
* Post pelvic radiotherapy.
* Vaginal/abdominal hysterectomy.
* Vaginal infection.
* Severe urinary tract infection.
* Uterine Prolapse

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — * Postmenopausal women (at least 12months after menstrual cessation), diagnosed with SUI by the gynecologist.
  * Their ages will range from 50-60 years old .
Enrollment: 60 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2024-08-20 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
• Revised urinary incontinence scale | 6 weeks
  : It is considered one of the tools which used to diagnose SUI. It takes the five best items which loaded on the urinary leakage. The items comprising this revised scale include urine leakage related to the feeling of urgency, urine leakage related to physical activity, coughing or sneezing, small amounts of urine leakage [drops]) as well as two items related to frequency and amount of incontinence Scoring is by simple summation and the range of the total score is between zero and 12(0= no incontinence , 1-2= slight incontinence , 3-6= moderate incontinence , 7-9= severe incontinence , 12= very severe incontinence)

SECONDARY OUTCOMES:
• Quality of Life Questionnaire (QOL) for stress urinary incontinence | 6 weeks
  : it has been developed to provide detailed information on how urinary incontinence affects patients' lives. It is a valid and reliable instrument for assessing QOL in women with voiding symptoms, including urinary incontinence. It includes questions that evaluate the distress and impact of urinary incontinence in three domains: avoidance and limiting behavior, social embarrassment and psychosocial impact